CLINICAL TRIAL: NCT01376063
Title: A Phase 1, Single-Center, One-Sequence, Open-Label Study to Investigate the Interaction Between FG-4592 and Rosiglitazone in Healthy Adult Subjects
Brief Title: Study to Investigate the Interaction Between FG-4592 and Rosiglitazone in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Robert Leong, MD., Medical Monitor, FibroGen, Inc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-037
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FG-4592 (Experimental)
  Interventions: Drug: FG-4592

INTERVENTIONS:
Drug: FG-4592 — FG-4592 on days 3,5,7,9
  Rosiglitazone maleate on days 1 and 9

SUMMARY:
The primary purpose of this study is to assess the effect of multiple doses of FG-4592 on the plasma pharmacokinetic of rosiglitazone in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males, 18 to 45 years
* Body weight ≥ 75 kg
* Good health
* Non-smoker
* Blood pressure not greater than 140/90 mm Hg

Exclusion Criteria:

* Positive for any of the following: Human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus antibody (anti-HCV Ab)
* Blood donation or significant blood loss within 60 days prior to Day 1
* Use of prescription and over the counter medications/herbal preparations is not allowed within 14 days prior to Day 1 and through treatment phase
* History or presence of alcoholism or drug abuse within 2 years prior to Day 1
* Consumption of alcohol within 7 days prior to Day 1 or during treatment phase
* Positive urine drug/alcohol testing at screening or check-in visit

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change in plasma concentration of Rosiglitazone | Day 1- Day 11

SECONDARY OUTCOMES:
Change in plasma concentration of Rosiglitazone metabolites | Day 3 - Day 11